CLINICAL TRIAL: NCT01803386
Title: Noninvasive Assessment of Neuromuscular Disease Using Electrical Impedance Myography
Status: Completed | Type: Observational
Sponsor: Skulpt, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: EIM-002-2011-4; 2R44NS070385-02A1 (NIH)
Record Dates: First submitted 2013-02-28; First posted 2013-03-04 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS)
Keywords: ALS; EIM
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- ALS Subjects: EIM measurements will be taken on two upper and two lower extremity muscles with several different electrode arrays. The ALSFRS-R will also be administered. Subcutaneous fat measurement will also be performed on all four muscles using skinfold calipers.
  Interventions: Device: EIM Measurements
- Healthy Subjects: EIM measurements will be taken on two upper and two lower extremity muscles with several different electrode arrays. Subcutaneous fat measurement will also be performed on all four muscles using skinfold calipers.
  Interventions: Device: EIM Measurements

INTERVENTIONS:
Device: EIM Measurements — EIM measurements are taken by applying saline to the skin and placing a sensor on patients' muscles that will record electrical activity. Electrical current is generated by this machine, but patients will not be able to feel it. The electrical activity recorded is returned to the machine and analyzed by a computer.
  Other Names: Electrical Impedance Myography Measurements

SUMMARY:
The purpose of this protocol is to test a new Electrical Impedance Myography (EIM) device and study its reliability and ability to differentiate ALS patients from healthy controls.

DETAILED DESCRIPTION:
Investigators will study 10 ALS patients and at least 10 age-matched healthy controls between the ages of 21 and 85 years old. For all subjects, EIM measurements will be performed on four muscles: two in the upper and two in the lower extremities, using 8 different EIM sensors. Measurements will be repeated one time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable or definite ALS by the El Escorial Criteria

Exclusion Criteria:

* History of superimposed generalized neuromuscular disease
* Primary lateral sclerosis or other atypical motor neuron disorders
* Forced vital capacity of less than 50%
* Presence of disease for greater than 5 years since symptom onset

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ALS Patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Muscle health as captured by EIM measurements | One time visit - Day 1
  EIM measurements will be performed with several electrode arrays at one visit per patient. The data captured from ALS and healthy subjects will be used to refine and finalize electrode array design development for the EIM system.

CONTACTS AND LOCATIONS:
Overall Officials: Erik Ensrud, MD, Principal Investigator — VA Boston Healthcare System
Locations (1):
- Convergence Medical Devices, Boston, Massachusetts, United States

REFERENCES:
- See also: Convergence Medical Devices Website — http://www.cmdevices.com